CLINICAL TRIAL: NCT05570084
Title: Randomised Controlled Trial on Silodosin Versus Tamsulosin for Medical Expulsive Treatment of Ureteral Stones Size 5-10mm in Chinese
Brief Title: Silodosin vs Tamsulosin as MET
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Princess Margaret Hospital, Hong Kong (Other Government)
Responsible Party: Principal Investigator, Ellen Yu, Research manager, Princess Margaret Hospital, Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KW/FR-19-075-(139-02)
Record Dates: First submitted 2022-09-28; First posted 2022-10-06 (Actual); Last update posted 2022-10-06 (Actual); Status verified 2022-10

CONDITIONS: Stone, Urinary
MeSH Terms: conditions — Urinary Calculi | interventions — silodosin; Tamsulosin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Tamsulosin (Active Comparator): 0.4mg daily for 4 weeks
  Interventions: Drug: Tamsulosin
- Silodosin (Experimental): 8mg daily for 4 weeks
  Interventions: Drug: Silodosin

INTERVENTIONS:
Drug: Silodosin — Cap silodosin for medical expulsion therapy
  Arms: Silodosin
Drug: Tamsulosin — Cap tamsulosin
  Arms: Tamsulosin

SUMMARY:
The spontaneous passage rate for ureteral stone less than 1cm causing acute ureteral obstruction is about 50%. Previous Cochrane review has concluded that alpha blocker is likely to increase stone passage rate, reduce time to stone passage, analgesic use and hospitalisations. The European Association of Urology Guideline also recommends giving alpha blockers as Medical Expulsive Therapy to patients with distal ureteric stones >5mm. However there is heterogeneity in different alpha blockers.

Silodosin is a recently introduced selective alpha blocker which has a much higher selectivity for the alpha-1-A receptor (17-fold compared with tamsulosin). From previous animal studies, ureteral contraction is mainly mediated by the alpha-1-A receptor, hence silodosin maybe more effective in increasing stone passage compared with tamsulosin.

Previous studies and meta-analysis has shown superiority of silodosin over tamsulosin on earlier stone passage and less pain. However, there is no data on Chinese population.

The investigators would like to compare the efficacy and side effect profile of Silodosin versus tamsulosin on improving stone passage rate and hence reduce rate of further intervention for stone clearance.

ELIGIBILITY:
Inclusion criteria:

* Presented with radio-opaque ureteric stone of size 5mm to 10mm on KUB
* Patients who can understand the study protocol and comply with the followup schedule

Exclusion criteria:

* Radiolucent stone
* Paper thin cortex
* Non-functioning kidney
* Renal insufficiency (serum creatinine greater than 1.8 mg/dl or 160umol/dL)
* Concurrent urosepsis
* Current [alpha]-blocker usage, Ca channel blocker, steroid
* Pregnancy
* Age < 18
* History of ureteral stricture
* History of ureteric stone treatment within 2 years
* Allergic reaction to the study medication
* Unable to Consent
* Patient on JJ stent or PCN drainage

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-05-31 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Stone free rate | FU at week 2
  Wet KUB for stone passage & RFT before FU (check 3/7 before the last FU)
Stone free rate | FU at week 4
  Wet KUB for stone passage & RFT before FU (check 3/7 before the last FU)

SECONDARY OUTCOMES:
Pain control | FU at week 2
  Use of analgesics and VAS pain scale (0-10)
Pain control | FU at week 4
  Use of analgesics and VAS pain scale (0-10)

CONTACTS AND LOCATIONS:
Locations (1):
- Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No